CLINICAL TRIAL: NCT04856592
Title: Clinical Outcomes of Intravascular Ultrasound-guided Stenting Using the Boston Scientific Vici® Venous Stent System in Treating Patients With Chronic Non-malignant Iliofemoral Vein Obstruction
Brief Title: Clinical Outcomes of IVUS-guided Stenting Using the Boston Scientific Vici® Venous Stent System in Treating Patients With Chronic Non-malignant Iliofemoral Vein Obstruction
Acronym: APAC VICI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study device VICI stent withdrawn from market
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2484
Record Dates: First submitted 2021-04-12; First posted 2021-04-23 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Chronic Venous Disorder; Venous Outflow Obstruction; Systemic Vein Outflow of Iliofemoral Vein

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- VICI Stent (Experimental)
  Interventions: Device: Boston Scientific Vici® Venous Stent System; Device: Boston Scientific Opticross 35 Peripheral Imaging Catheter (OC35 catheter)

INTERVENTIONS:
Device: Boston Scientific Vici® Venous Stent System — The Vici Venous Stent System comprises two components: the implantable endoprosthesis and its stent delivery system, a 9F over-the-wire system available in a 100cm length and compatible with 0.035in (0.89mm) guidewires
Device: Boston Scientific Opticross 35 Peripheral Imaging Catheter (OC35 catheter) — The Opticross 35 catheter is designed for use with a guidewire measuring ≤0.035 in (0.89 mm) in diameter and an introducer sheath of 8F (2.67 mm) or larger. The working length of OC35 catheter is 105 cm.

SUMMARY:
The APAC VICI Study is a prospective, non-randomized, multicenter, single-arm study. The purpose of this study is to evaluate the clinical results of using the Boston Scientifc's Vici Venous Stent (Vici stent) to treat significant blockage in the iliofemoral veins under the guidance of intravascular ultrasound (IVUS) in ethnic Chinese patient population. The study will assess the safety and effectiveness of Vici stent implanted under the guidance of the Boston Scientific's IVUS technology (by using Opticross 35 catheter) for treating adult ethnic Chinese patients with symptomatic chronic venous obstruction in the iliofemoral veins.

During the trial, anticoagulant or antiplatlet therapy will be administered for 6 - 12 months post index procedure. Ongoing dynamic data safety monitoring will be performed throughout the trial to minimize subject risk. All enrolled subjects receiving the Vici stent treatment will be followed for 24 months post index procedure.

ELIGIBILITY:
Key Inclusion Criteria:

1. Ethnic Chinese subjects of age ≥ 18 years (or meet age requirements per local law)
2. Subjects willing to provide written informed consent prior to the study and AND willing to comply with all follow-up evaluations at the specified times
3. Subjects with presence of unilateral, clinically significant, chronic non-malignant obstruction of the common femoral vein, external iliac vein, common iliac vein, or any combination thereof, defined as a > 50% reduction in target vessel lumen diameter measured by venogram and/or IVUS during procedure
4. Clinically significant venous obstruction defined as meeting at least one of the following clinical indicators:

   * Clinical severity class of CEAP classification ≥ 3
   * rVCSS Pain Score ≥ 2
5. Negative pregnancy test in female subjects of potential child-bearing
6. Intention to stent the target lesion only with the Vici Stent(s)

Key Exclusion Criteria:

Pre-Procedural EC--

1. Subjects with presence or history of clinically significant pulmonary emboli within 6 months prior to enrollment.
2. Subjects with venous obstruction that extends into the inferior vena cava
3. Subjects with contralateral disease of the common femoral vein, external iliac vein, common iliac vein, or any combination thereof with planned treatment within 30 days after enrollment
4. Subjects with a life expectancy < 12 months
5. Female of childbearing potential who is pregnant or plans to become pregnant during the duration of the clinical study (Note: subjects who plan to become pregnant after 12-month follow-up visit may be included in the trial at the discretion of treating physician)
6. A. Subjects with uncontrolled or active coagulopathy OR

   B. Subjects with known uncorrectable bleeding diathesis with the following definitions:
   * Uncorrected INR ≥ 2.0 or aPTT ≥ 1.5X normal local lab value
   * Platelet count < 80,000
7. Subjects with uncorrected hemoglobin of ≤ 9 g/dL
8. Subjects with an estimated glomerular filtration rate (eGFR) < 30 mL/min. In patients with diabetes mellitus, eGFR < 45 mL/min.
9. Subjects have known hypersensitivity to nickel or titanium
10. Subjects have contrast agent allergy that cannot be managed adequately with pre-medication
11. Subjects will have intended concurrent thrombolysis or thrombectomy procedure OR intended or planned (within 30 days) adjuvant procedure such as creation of temporary AV fistula, placement of IVC filter, endovenectomy or saphenous vein ablation
12. Subjects currently participating in another drug or device clinical trial (participation in observational studies is acceptable)
13. Subjects judged to be a poor candidate by the primary investigator
14. Subjects who have had any prior surgical or endovascular intervention of the target vessel

Intra-Procedural:

1. Subjects in whom the lesions cannot be traversed with a guide wire
2. Subjects where the obstruction extends into the inferior vena cava or below the level of the lesser trochanter
3. Subjects whose vein diameters are not within limits stated in the Instructions for Use of study device as determined by venogram and/or IVUS
4. Subjects who do not meet the venogram or IVUS binary stenosis by the definition above (IC3), as determined by the treating physician
5. Subjects who are judged by treating physician to have a lesion that prevents completed inflation of a balloon dilation catheter or proper placement of the stent or the stent delivery system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary patency rate at 12 months post index procedure | 12 month
  Defined as freedom from occlusion by thrombosis AND freedom from surgical or endovascular intervention on target vessel which are found to have restenosis or stent occlusion to maintain patency AND freedom from in-stent stenosis more than 50% by DUS.
Major Adverse Events within 30 days post index procedure | 30 days
  The composite endpoint of below major adverse events (MAE) adjudicated by the Clinical Events Committee (CEC) within 30 days post index procedure:
  * Device or procedure-related death
  * Device or procedure-related bleeding at the target vessel and/or the target lesion or at the access site requiring surgical or endovascular intervention or blood transfusion ≥ 2 units
  * Device or procedure-related arterial or venous injury occurring in the target vessel segment and/or target lesion or at the access site requiring surgical or endovascular intervention
  * Device or procedure related acute DVT outside of the target vein segment
  * Clinically significant pulmonary embolism defined as being symptomatic with chest pain, hemoptysis, dyspnea, hypoxia etc… AND be documented on CT
  * Stent embolization
  * Stent thrombosis

IPD SHARING:
Plan to Share IPD: Undecided